CLINICAL TRIAL: NCT05722678
Title: Study and Analysis on the Characteristics of Intestinal Microorganisms and Serum Metabolites in Patients With Acute Pancreatitis Complicated With COVID-19
Brief Title: Study and Analysis of Acute Pancreatitis Complicated With COVID-19
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yuansong Sun (Other)
Collaborators: Anhui Medical University (Other); Nanjing University (Other)
Responsible Party: Sponsor-Investigator, Yuansong Sun, attending doctor, The Second Hospital of Anhui Medical University
Organization: The Second Hospital of Anhui Medical University (Other)
Other Study IDs: KY20221224
Record Dates: First submitted 2023-01-29; First posted 2023-02-10 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Acute Pancreatitis; 2019 Novel Coronavirus Infection
Keywords: Novel coronavirus infection; Acute pancreatitis; Intestinal flora; Serum metabolism
MeSH Terms: conditions — Pancreatitis; COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study was to explore the complex relationship between changes in the intestinal microbiome and serum metabolites in patients with novel coronavirus infection and acute pancreatitis. The main questions it aims to answer are:

Question 1: The changes of intestinal microbiota and serum metabolites in patients with novel coronavirus infection and acute pancreatitis.

Question 2: The relationship between the changes in the intestinal microbiome and serum metabolites.

Participants will be recruited according to certain criteria. The investigators plan to recruit 4 groups of 30 volunteers, 120 volunteers in total. It is divided into (a) AP patients without COVID-19 (normal group) (b) AP patients with COVID-19 (treatment group) (c) patients with COVID-19 infection (control group) (d) normal healthy people. The basic information of subjects, including age, sex, address, and enrollment time, was collected after enrollment. After completing the relevant preparations, start the experiment. First of all, the sample collection and detection. Blood samples were taken from 2-3ml of blood (biochemical tube) after admission or in the morning of the next day, centrifuged at 3000 rpm for 3 minutes, and stored at -80℃ within 1 hour after taking the serum; Fecal samples are stool samples retained after admission and before antibiotic use. Fecal samples need to be stored at -20℃ within one hour after collection and transferred to -80℃within 24 hours. After the retention of samples, the retained stool samples shall be tested for bacterial flora, and the blood samples shall be tested for serum metabolomics. After the test, the investigators will use the statistical software SPSS 22.0 for statistical analysis. At the same time, in order to determine the correlation between intestinal flora and clinical parameters, the investigators will use Permutation analysis of variance (PERMANOVA) to process the data.

DETAILED DESCRIPTION:
Acute pancreatitis (AP) is a common gastrointestinal disease. In recent years, the hospitalization rate and related costs of AP have increased significantly. About 15% - 20% of patients will develop acute severe pancreatitis, namely SAP. SAP is a serious abdominal disease with many complications and high mortality. The global average annual incidence rate is about 6.75 cases/100000 people. Systemic inflammatory response syndrome (SIRS), multiple organ dysfunction syndrome (MODS), and sepsis are often associated with it. SIRS and MODS may be caused by the release of inflammatory cytokines in the early stage of AP, and intestinal dysfunction and pancreatic necrosis in the later stage. Some studies have shown that 59% of AP patients are accompanied by intestinal barrier injury, and increased permeability of intestinal mucosa, resulting in intestinal bacterial translocation, pancreatic tissue necrosis and infection, and multiple organ dysfunction syndrome. Most of the bacteria causing necrotic infection of pancreatic tissue to come from intestinal flora, such as Escherichia coli and Enterococcus. Therefore, intestinal flora may play an important role in the occurrence and development of AP.

As the largest organ of the human body, the gastrointestinal tract provides a broad colonization surface for biological flora. Intestinal bacteria present in the human gastrointestinal tract are essential components for the development of the mucosal immune system, the promotion of food digestion and absorption, and the regulation of glucose metabolism. In addition, it also has the function of protecting the intestinal barrier and mediating host immunity and metabolism. The host and microbe reach the micro-ecological balance in the state of health, which is called internal environment stability, and the host maintains normal physiological functions. However, external factors (such as infection, toxin, diet change, disease, etc.) may change or destroy the balance between them, and the disorder of intestinal flora will in turn induce or accelerate the disease's progress. As one of the research hotspots in recent years, the imbalance of intestinal flora has always attracted people's attention. The current study found that the ecological imbalance of intestinal microbiota during AP was defined as the decrease of intestinal microbial diversity and the change of the balance between symbiotic microbiota and pathogenic microbiota. The change of intestinal flora occurred in the early stage of AP, which may be involved in the aggravation of the disease. Not only that but also early intestinal flora disorder was found in SAP research. In addition to intestinal bacteria, their metabolites such as short-chain fatty acids (SCFAs) also affect the progress of AP. Moreover, more and more studies have found that changes in intestinal flora during the development of AP may be related to the severity of the disease. In the process of AP occurrence and development, the abnormal secretion of trypsin and the destruction of pancreatic structure leads to the abnormal secretion of the pancreas, which can cause changes in intestinal homeostasis and intestinal flora. In addition, the study also found that intestinal microbiota is an important medium during AP, and its imbalance is closely related to the severity of AP. At present, many experimental data have shown that the diversity of intestinal microorganisms and the relative abundance of specific bacterial groups have changed during the AP process.

Based on the relationship between intestinal flora imbalance and the occurrence and development of AP, the possible mechanisms of intestinal microbial imbalance in AP are mainly as follows: (1) intestinal motility disorder: gastrointestinal motility disorder often exists in AP and plays a role in disease progression. Intestinal motility disorder can also lead to the accumulation of harmful substances and inhibit the growth of probiotics. (2) Ischemia-reperfusion injury (IRI): pro-inflammatory cytokines such as TNF- α during AP, the release of insulin can cause intestinal mucosal IRI and disrupt intestinal microcirculation. One of the main causes of intestinal microcirculation damage is the destruction of sugar calyx. (3) Oxidative stress: severe oxidative stress and intestinal-activated caspase-3 pathway was found during AP. Oxidative stress not only accelerates the disorder of intestinal barrier function but also participates in the disorder of intestinal microbiota. (4) Immune dysfunction: intestinal immunosuppression can be observed in the early stage of acute pancreatitis, which is related to the damage of the clearance of proliferative pathogens.

In AP, the change of intestinal microflora is closely related to its occurrence and development, and the metabolites of intestinal microflora will also affect the serum metabolic indicators of AP patients. Intestinal microflora has high metabolic activity and can transform host sources and dietary components into different metabolites. Some metabolites are beneficial and some are harmful. Metabolites beneficial to the host include lactic acid, bile acid (BA), SCFA, and bacteriocin. These substances are generally considered antibacterial factors and play a key role in the prevention of pathogenic infection. In addition, there are also related intestinal flora and several specific products produced that may have a certain impact on SAP. In human intestines, bifidobacteria and lactobacillus are probiotics that can stimulate anti-tumor properties and immunity. The main products of bifidobacterium metabolism are lactic acid and acetic acid, which reduce the pH value in the intestine and inhibit the growth of harmful microorganisms. This mechanism is particularly evident in the cecum and ascending colon.

At present, the continuous pandemic of coronavirus disease (COVID-19) in 2019 caused by severe acute respiratory syndrome coronavirus type 2 (SARS-CoV-2) poses a serious threat to global public health, and millions of people in more and more countries are at risk. This pandemic has not only affected the medical system but also affected the global socioeconomic balance. COVID-19 was soon designated as a global pandemic by the World Health Organization, because as of January 2021, there were about 98 million confirmed cases and about 2 million confirmed deaths. Nevertheless, since the outbreak of COVID-19, our understanding of it has increased significantly, and a variety of treatment methods and drug interventions have been tested or are currently being developed to reduce its risk factors. Recently, some candidate vaccines have shown about 95% clinical efficacy and are currently being approved for emergency use in different countries. Therefore, vaccination as one of the effective means of protection is worth promoting worldwide. Some studies have confirmed that several intestinal microflorae have the potential to improve the immune response and reduce adverse events after COVID-19 vaccination and that intestinal microflora has the potential to supplement the effectiveness of the vaccine. Combined with several recent studies, intestinal flora plays a key role in regulating the immune response to vaccination and is related to the severity of COVID-19 patients. However, the comprehensive evaluation of host response, especially the role of intestinal flora in antibody production, is limited. Therefore, the specific role of intestinal flora in the development of COVID-19 needs further study.

The composition of intestinal microflora and the severity of acute infection (including COVID-19) have a two-way relationship with the lung, which is called the "gut-lung axis". Intestinal ecological imbalance, that is, the emergence of viral pathological organisms, changes the signal transduction of intestinal epithelial cells and produces proinflammatory reactions, which can lead to impaired immune response and make COVID-19 patients vulnerable to serious diseases. A variety of inflammatory and infectious diseases are associated with symbiotic disorders. Several studies have shown that the stool virus shedding of COVID-19 patients will continue for a long time after the respiratory symptoms subside. This shows that the gastrointestinal tract is the site of virus replication, and has caused concern about fecal and oral transmission. This was further confirmed by a small study of 30 COVID-19 patients. The study showed that the decrease in biological diversity increased along with the increase of opportunistic bacteria, including Streptococcus, Rochella, Verona, Clostridium erysipelas, and actinomycetes. The abundance of fecal bacteria, Clostridium mycobacterium and Clostridium hartwickii was associated with severe COVID-19 disease. The abundance of beneficial Bacteroides and Alisma orientalis was negatively correlated with the severity of the disease. Many studies have explored the relationship between intestinal ecological disorders, severe COVID-19, and elevated inflammatory markers. Bacteroides Donovan and Akermann myxophila and IL-1 β、 IL-6 are positively correlated with CXCL8. Similarly, IL10, TNF- α, and chemokines (such as CXCL10 and CCL2) are negatively correlated with beneficial microbiota (such as Bifidobacterium adolescents, Eubacterium rectum and Faecalis procterii), which maintain a low level in fecal samples collected one month after the disease. In another study involving a small group of COVID-19 patients, butyric acid producers (for example, Fecal Procter, Clostridium butyricum, Clostridium parvum, and Eubacterium rectum) were significantly reduced, and conditional pathogens such as Enterococcus and Enterobacteriaceae were abundant in severe patients with adverse outcomes. Changes in intestinal microflora were observed in children with acute and non-acute Kawasaki disease, which further suggested that MISC in SARS-CoV-2 might be associated with ecological disorders. Limited studies on patients with COVID-19 have shown intestinal ecological disorders. A small report at the beginning of the pandemic showed that the levels of lactobacilli and bifidobacteria in COVID-19 patients were low. Zuo et al. showed that COVID-19 virus RNA in the feces of almost half of the sampled patients was positive, which lasted for a long time after the respiratory tract was cleared. In addition, the authors found that patients with viral RNA had higher levels of opportunistic pathogens. To better clarify the role of probiotics in the treatment of COVID-19, several studies are currently underway. The clear recommendations on probiotics and COVID-19 treatment still need further evidence, although there are biological rationality and reasons to hope that they may play a beneficial role.

In the current era of the continuous prevalence of COVID-19, many patients are faced with COVID-19 infection and AP at the same time, which poses new challenges to the diagnosis and treatment of clinicians. Based on the key role of intestinal flora imbalance in AP and COVID-19 infection and the unique advantages of metabonomics in the diagnosis and prognosis of infectious diseases. Therefore, our research is based on the fact that the imbalance of intestinal flora plays an important role in the development of COVID-19 infection and AP while considering the impact of intestinal flora and its metabolites on the serological indicators of patients. The purpose of this study was to explore the complex relationship between the changes in the intestinal microbiome and serum metabolite in patients with novel coronavirus infection and acute pancreatitis, hoping to provide help for clinical diagnosis and treatment of patients with novel coronavirus infection and acute pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

* voluntary enrollment and consent to retain biological samples for research, and signing the informed consent form;
* In recent 2 days, it was confirmed that COVID-19 with acute pancreatitis, and the diagnosis was clear. Among them, the diagnostic standard of acute pancreatitis is the International Consensus on Acute Pancreatitis, revised in Atlanta in 2012;
* Subjects did not receive treatment before enrollment

Exclusion Criteria:

* have received treatment before hospitalization;
* The patient has a malignant tumor, infectious disease or allergic disease;
* Combined with immune diseases or other acute and chronic inflammatory diseases;
* The patient was diagnosed with intestinal dysfunction recently;
* The patient has communication or cognitive impairment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The investigators plan to recruit 4 groups of 30 volunteers, 120 volunteers in total. It is divided into (a) AP patients without COVID-19 (normal group) (b) AP patients with COVID-19 (treatment group) (c) patients with COVID-19 (control group) (d) normal healthy people.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-02-15 (Estimated); Primary Completion 2023-06-12 (Estimated); Study Completion 2023-06-12 (Estimated)

PRIMARY OUTCOMES:
Changes of intestinal microflora abundance in feces | through study completion, an average of 6 months
  The relationship between the abundance of each common bacteria in the feces of patients in the experimental group and the change of the normal control group
Changes of metabolic indexes in blood samples | through study completion, an average of 6 months
  The change relationship between the common laboratory metabolic blood indicators in the blood of patients in the experimental group and the normal control group

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers

REFERENCES:
- [Background] Portelli M, Jones CD. Severe acute pancreatitis: pathogenesis, diagnosis and surgical management. Hepatobiliary Pancreat Dis Int. 2017 Apr;16(2):155-159. doi: 10.1016/s1499-3872(16)60163-7. PMID 28381378
- [Background] Schietroma M, Pessia B, Carlei F, Mariani P, Sista F, Amicucci G. Intestinal permeability and systemic endotoxemia in patients with acute pancreatitis. Ann Ital Chir. 2016;87:138-44. PMID 27179282
- [Background] Gao R, Wu C, Zhu Y, Kong C, Zhu Y, Gao Y, Zhang X, Yang R, Zhong H, Xiong X, Chen C, Xu Q, Qin H. Integrated Analysis of Colorectal Cancer Reveals Cross-Cohort Gut Microbial Signatures and Associated Serum Metabolites. Gastroenterology. 2022 Oct;163(4):1024-1037.e9. doi: 10.1053/j.gastro.2022.06.069. Epub 2022 Jul 1. PMID 35788345
- [Background] Li XY, He C, Zhu Y, Lu NH. Role of gut microbiota on intestinal barrier function in acute pancreatitis. World J Gastroenterol. 2020 May 14;26(18):2187-2193. doi: 10.3748/wjg.v26.i18.2187. PMID 32476785
- [Background] Majumder J, Minko T. Recent Developments on Therapeutic and Diagnostic Approaches for COVID-19. AAPS J. 2021 Jan 5;23(1):14. doi: 10.1208/s12248-020-00532-2. PMID 33400058
- [Background] Chilamakuri R, Agarwal S. COVID-19: Characteristics and Therapeutics. Cells. 2021 Jan 21;10(2):206. doi: 10.3390/cells10020206. PMID 33494237
- [Background] Yoshikawa T, Watanabe T, Kamata K, Hara A, Minaga K, Kudo M. Intestinal Dysbiosis and Autoimmune Pancreatitis. Front Immunol. 2021 Mar 23;12:621532. doi: 10.3389/fimmu.2021.621532. eCollection 2021. PMID 33833754
- [Background] Wang Z, Li F, Liu J, Luo Y, Guo H, Yang Q, Xu C, Ma S, Chen H. Intestinal Microbiota - An Unmissable Bridge to Severe Acute Pancreatitis-Associated Acute Lung Injury. Front Immunol. 2022 Jun 14;13:913178. doi: 10.3389/fimmu.2022.913178. eCollection 2022. PMID 35774796
- [Background] Zhu Y, Mei Q, Fu Y, Zeng Y. Alteration of gut microbiota in acute pancreatitis and associated therapeutic strategies. Biomed Pharmacother. 2021 Sep;141:111850. doi: 10.1016/j.biopha.2021.111850. Epub 2021 Jun 30. PMID 34214727
- [Background] Ye S, Si C, Deng J, Chen X, Kong L, Zhou X, Wang W. Understanding the Effects of Metabolites on the Gut Microbiome and Severe Acute Pancreatitis. Biomed Res Int. 2021 Oct 19;2021:1516855. doi: 10.1155/2021/1516855. eCollection 2021. PMID 34712726
- [Background] Hasan MR, Suleiman M, Perez-Lopez A. Metabolomics in the Diagnosis and Prognosis of COVID-19. Front Genet. 2021 Jul 23;12:721556. doi: 10.3389/fgene.2021.721556. eCollection 2021. PMID 34367265
- [Background] Liu R, Hong J, Xu X, Feng Q, Zhang D, Gu Y, Shi J, Zhao S, Liu W, Wang X, Xia H, Liu Z, Cui B, Liang P, Xi L, Jin J, Ying X, Wang X, Zhao X, Li W, Jia H, Lan Z, Li F, Wang R, Sun Y, Yang M, Shen Y, Jie Z, Li J, Chen X, Zhong H, Xie H, Zhang Y, Gu W, Deng X, Shen B, Xu X, Yang H, Xu G, Bi Y, Lai S, Wang J, Qi L, Madsen L, Wang J, Ning G, Kristiansen K, Wang W. Gut microbiome and serum metabolome alterations in obesity and after weight-loss intervention. Nat Med. 2017 Jul;23(7):859-868. doi: 10.1038/nm.4358. Epub 2017 Jun 19. PMID 28628112
- [Background] Han M, Huang Y, Gui H, Xiao Y, He M, Liu J, Cao X, Zheng M, Lu M, Jia W, Li H, Wang X, Zhang N, Kong SA, Liu X, Wu Y, Wu F, Huang S. Dynamic changes in host immune system and gut microbiota are associated with the production of SARS-CoV-2 antibodies. Gut. 2023 Oct;72(10):1996-1999. doi: 10.1136/gutjnl-2022-327561. Epub 2022 Oct 7. No abstract available. PMID 36207022